CLINICAL TRIAL: NCT02955342
Title: Back and Neck Pain in Adolescence: A Prospective Cohort Study Using a German Version of the Young Spine Questionnaire
Brief Title: Back and Neck Pain in Adolescence
Acronym: Youngback
Status: Completed | Type: Observational
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-00568
Record Dates: First submitted 2016-10-06; First posted 2016-11-04 (Estimated); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To validate the German version of the Young Spine Questionnaire (G-YSQ) and to study back and neck pain in adolescents between 10 and 16 years during one year by means of G-YSQ.

DETAILED DESCRIPTION:
In two settings (school, clinics) back and neck pain of 10 to 16 years old adolescents will be assessed by the German Version of the Young Spine Questionnaire at 6 points in time during one year.

Validity, reliability and responsiveness of the G-YSQ will be determined and the development of back and neck pain within a year will be described.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 16 years old

Exclusion Criteria:

* younger than 10, older than 16

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents between 10 and 16 years with and without back and neck pain.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-07 (Actual)

PRIMARY OUTCOMES:
Changes in a German Version of the Young Spine Questionnaire | change from baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry K Humphreys, Professor, Study Director — Balgrist University Hospital
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lauridsen HH, Hestbaek L. Development of the young spine questionnaire. BMC Musculoskelet Disord. 2013 Jun 12;14:185. doi: 10.1186/1471-2474-14-185. PMID 23758965
- [Background] Wirth B, Knecht C, Humphreys K. Spine Day 2012: spinal pain in Swiss school children- epidemiology and risk factors. BMC Pediatr. 2013 Oct 5;13:159. doi: 10.1186/1471-2431-13-159. PMID 24094041
- [Background] Wirth B, Humphreys BK. Pain characteristics of adolescent spinal pain. BMC Pediatr. 2015 Apr 17;15:42. doi: 10.1186/s12887-015-0344-5. PMID 25886130
- [Derived] Nyiro L, Potthoff T, Siegenthaler MH, Riner F, Schweinhardt P, Wirth B. Translation and validation of the German version of the Young Spine Questionnaire. BMC Pediatr. 2021 Aug 24;21(1):359. doi: 10.1186/s12887-021-02804-y. PMID 34429090